CLINICAL TRIAL: NCT01593189
Title: A Randomized Efficacy Trial of the Kids in Transition to School (KITS) Program for Children With Developmental Disabilities and Behavioral Problems
Brief Title: Efficacy Trial of the Kids in Transition to School (KITS) Program for Children With Developmental Disabilities and Behavioral Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Social Learning Center (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Katherine C. Pears, Research Scientist, Oregon Social Learning Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R324A080026
Record Dates: First submitted 2012-05-02; First posted 2012-05-08 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: School Readiness
Keywords: developmental disabilities; school readiness; literacy; social emotional skills; self regulation; caregiver involvement
MeSH Terms: conditions — Developmental Disabilities; Literacy; Self-Control

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- KITS Program (Experimental): The KITS intervention consists of: (a) child school readiness play groups to facilitate the development of self-regulatory, social, and early literacy skills (2 times per week in summer, 1 times per week in the fall); and (b) a bi-monthly psychoeducational support group to promote parent involvement in the child's early literacy and schooling and the use of effective parenting techniques
  Interventions: Behavioral: KITS Program
- Services as usual (No Intervention): Families continued to receive any services that they had been receiving in the community.

INTERVENTIONS:
Behavioral: KITS Program — This is a 4-month psychosocial intervention for children with developmental disabilities and behavior problems who are entering kindergarten and their caregivers. The intervention begins in the summer before kindergarten. The KITS intervention consists of: (a) child school readiness play groups to facilitate the development of self-regulatory, social, and early literacy skills (2 times per week in summer, 1 times per week in the fall); and (b) a bi-monthly psychoeducational support group to promote parent involvement in the child's early literacy and schooling and the use of effective parenting techniques
  Other Names: Kids in Transition to School (KITS) Program
  Arms: KITS Program

SUMMARY:
This study focuses on children entering kindergarten with co-occurring developmental disabilities and behavior problems, a population especially likely to have low levels of school readiness. Prior research has shown that children with developmental disabilities are at risk for academic difficulties. Behavioral and social problems are likely to interfere with school adjustment. The investigators hypothesize that children who receive the intervention will show better school readiness and school adjustment outcomes.

DETAILED DESCRIPTION:
Purpose: This project is a randomized efficacy trial of KITS, an intervention to enhance social-emotional and early literacy domains of school readiness in children with co-occurring developmental disabilities and behavior problems who are entering kindergarten.

Setting: The setting for the intervention will be playgroups and parent support groups conducted in center-based classrooms during the summer before and the first 2 months of kindergarten.

Population: This study involves the recruitment of 200 children with co-occurring developmental disabilities and behavioral problems who are entering kindergarten in the fall (four yearly cohorts of 50 children each). The children will be recruited from the Lane County, Oregon, public agency responsible for early childhood special education services.

Intervention: KITS is a short-term, intensive program timed to occur during the transition to kindergarten-a critical developmental milestone with far-reaching effects on school outcomes. The KITS curriculum focuses on the social-emotional and early literacy skills shown to be essential for success in kindergarten and on contextual characteristics (i.e., parent involvement in early literacy and positive parenting) to support and promote these skills. KITS features 24 curriculum-based school readiness playgroups to facilitate the development of self-regulatory, social, and early literacy skills (twice weekly in the summer before kindergarten and once weekly September-October) and 7 psychoeducational parent groups focused on parent involvement in early literacy and positive parenting practices (every 2 weeks June-October).

Research Design and Methods: Children will be randomly assigned to the KITS intervention condition or a services-as-usual comparison group and assessed at four intervals: spring prior to kindergarten, immediately prior to kindergarten entry, kindergarten fall, and kindergarten spring. One hundred fifty of the children will also be assessed in the spring of first grade. KITS children will receive the intervention as described above.

Control condition: Children in the comparison group will receive any ECSE or other services that they would typically receive. These will be assessed at each data collection point.

Key measures: Multimethod, multiagent outcome measures will include the following: direct assessments of the child's social-emotional and early literacy skills prior to kindergarten and social-emotional functioning and literacy skills during kindergarten and first grade; parent and teacher reports on children's characteristics, parent involvement in early literacy and school, and parenting practices; and direct classroom observations of children's academic engaged time and social behaviors during unstructured school time.

Data-analytic strategies: Analyses will employ variable-based (e.g., ANOVA and regression) and person-based (e.g., latent growth curve modeling) approaches. SEM will be used to test how changes in hypothesized mediators affect outcomes and how outcomes vary depending on level of hypothesized moderators.

ELIGIBILITY:
Inclusion Criteria:

* Received early childhood special education services
* Judged to have behavioral problems that would interfere with the transition to kindergarten
* Entering kindergarten in the fall of the year in which recruited into the study

Exclusion Criteria:

* Mono-lingual Spanish speaker
* Severe visual, hearing or physical impairment that would prevent the child from completing the assessment tasks or participating in the intervention

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 209 (Actual)
Dates: Start 2008-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in caregiver involvement from baseline to kindergarten entry | pre-intervention (baseline), pre-kindergarten ( approximately 2 months post-baseline)
  Caregiver reported involvement in early literacy activities and beliefs about the importance of various literacy skills for kindergarten
Change in early literacy skills from baseline to kindergarten entry | pre-intervention (baseline), pre-kindergarten ( approximately 2 months post-baseline)
  Standardized measures of early literacy skills including letter naming, phonological awareness and understanding of concepts about print
Change in social skills from baseline to kindergarten entry | pre-intervention (baseline), pre-kindergarten ( approximately 2 months post-baseline)
  Standardized direct assessments of the child's responses to social situations as well as parent responses to standardized questionnaires on children's social skills
Change in regulatory skills from baseline to kindergarten entry | pre-intervention (baseline), pre-kindergarten ( approximately 2 months post-baseline)
  Standardized direct assessment of the children's executive function skills as well as parent report on standardized questionnaires used to assess emotion and behavior regulation

SECONDARY OUTCOMES:
Longitudinal academic achievement across grade levels | post-kindergarten (approximately 1 year post-baseline), post 1st grade (approximately 2 years post-baseline)
  Standardized direct assessments of child achievement in reading and math as well as parent and teacher report on standardized measures of child achievement.
Longitudinal social competence across grade levels | post-kindergarten (approximately 1 year post-baseline), post 1st grade (approximately 2 years post-baseline)
  Standardized direct child assessments of responses to peer situations as well as child report on standardized questionnaires about social functioning at school and parent and teacher reports of child social functioning on standardized questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Social Learning Center, Eugene, Oregon, United States

REFERENCES:
- [Background] Pears KC, Fisher PA, Heywood CV, Bronz KD. Promoting school readiness in foster children. In: Saracho ON, Spodek B, eds. Contemporary Perspectives on Social Learning in Early Childhood Education Greenwich, CT: Information Age Publishing; 2007:173-198.
- [Background] Pears KC, Kim HK, Healey CV, Yoerger K, Fisher PA. Improving child self-regulation and parenting in families of pre-kindergarten children with developmental disabilities and behavioral difficulties. Prev Sci. 2015 Feb;16(2):222-32. doi: 10.1007/s11121-014-0482-2. PMID 24676874
- See also: Oregon Social Learning Center web site — http://www.oslc.org